CLINICAL TRIAL: NCT06704386
Title: Life Beyond Pain and Loss: A Comperative Analysis of Quality of Life in Chronic Pain and Amputee Patients
Brief Title: Chronic Pain and Amputation: A Quality of Life Comparison
Status: Active, not recruiting | Type: Observational
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Gamze Gul Gulec, Doctor, Baskent University
Other Study IDs: 24/191
Record Dates: First submitted 2024-11-07; First posted 2024-11-26 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Amputation
Keywords: Amputation; quality of life; chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Patients with amputations: Patients with amputation who are over 18 years of age, have sufficient Turkish reading and comprehension skills, and have experienced at least one year since the amputation, excluding those with congenital amputations or chronic pain.
- Patients with Chronic Pain: Patients with chronic pain who are over 18 years of age, have experienced pain for more than 3 months, and possess sufficient Turkish reading and comprehension skills.

SUMMARY:
The aim of this observational, cross-sectional study is to investigate and compare the impact of chronic pain and amputation on patients' quality of life. By excluding individuals with conditions that might influence quality of life, the study seeks to provide insights into how these two conditions affect physical and emotional well-being. Statistical methods will be employed to analyze the data. The primary research questions are as follows:

Is the quality of life of individuals with chronic pain lower than that of those with an amputation? Is the quality of life of individuals with chronic pain higher than that of those with an amputation? Is the quality of life of individuals with chronic pain similar to that of those with an amputation?

DETAILED DESCRIPTION:
Chronic pain is a common, complex, and distressing public health issue that significantly impacts both individuals and society, affecting more than 30% of the global population. Each year, 1 in 10 people develop chronic pain, making it one of the leading causes of disability worldwide. It is also one of the primary reasons patients seek medical care. The economic burden of chronic pain rivals that of cancer and cardiovascular diseases. Chronic pain is a multidimensional health problem, influencing every aspect of patients' lives. It contributes to loss of function and is accompanied by physical, emotional, cognitive, psychosocial, and motivational challenges. Additionally, it is associated with reduced activity levels, impaired functionality, and a significant decline in quality of life.

Amputation, on the other hand, is a major trauma that results in profound changes to body structure and function, substantially affecting an individual's quality of life, both socially and professionally. It creates barriers to reintegration into work and social life, limiting active participation in society. Amputation has far-reaching impacts on quality of life, including body image concerns, loss of a sense of integrity, decreased self-esteem, a distorted body image, feelings of emptiness and worthlessness, difficulties with social adjustment, reduced sexual activity, anxiety, depression, social discomfort, and challenges in relationships and marriage.

Health is defined as a state of complete physical, social, and spiritual well-being. Both chronic pain and amputation impair individuals' health status due to limitations in physical and social functioning, mental health challenges, pain, and reduced health-related quality of life. While numerous studies have explored the quality of life associated with each condition, no study has directly compared the quality of life between individuals with chronic pain and those who have undergone amputation.

The aim of this study is to compare the quality of life of individuals with chronic pain to that of amputees, providing valuable insights into the unique and overlapping challenges faced by these patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old or older
* Having adequate Turkish reading and understanding skills
* Having pain for more than 3 months (for patients with chronic pain)
* At least 1 year having passed since the amputation (for patients with amputatiton)

Exclusion Criteria:

* Having additional diseases such as stroke, multiple sclerosis, arthrosis, and psychiatric disorders, which could limit their physical and emotional status, so the quality of life
* Pregnancy Experiencing pain due to malignancy (for patients with chronic pain)
* Congenital amputation and chronic pain (for patients with amputatition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain and amputations will be recruited from the outpatient clinic of Physical Medicine and Rehabilitation Department
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Short Form -36 (SF-36) | From November 14 to December 17
  The SF-36 is one of the most widely used generic tools for measuring quality of life.This scale evaluates eight health dimensions across 36 items: physical function, role limitations (due to physical and emotional problems), social function, mental health, vitality (energy), pain, and general health perception.
  The SF-36 offers several advantages, including its ability to assess both the positive and negative aspects of a health condition in just five minutes.It also demonstrates superior sensitivity in detecting subtle changes in disability compared to other scales. Instead of providing a single score, the SF-36 generates separate scores for each subscale, ranging from 0 to 100. A score of 100 indicates excellent health, while a score of 0 reflects poor health.
  It has been validated and found reliable in Turkish and is recommended for use across all physical disease groups to assess quality of life comprehensively.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Adana Dr Turgut Noyan Research and Training Center, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No